CLINICAL TRIAL: NCT03881410
Title: The Efficacy of Shear-wave Elastography-guided Aspiration and Biopsy for Diagnosis in Lung Tumor: a Randomized Controlled Trial
Brief Title: The Efficacy of Shear-wave Elastography-guided Aspiration and Biopsy for Diagnosis in Lung Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201812180RINA
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2023-07

CONDITIONS: Lung Tumor
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shear-wave elastography-guided (Experimental): Shear-wave elastography-guided bipsy
  Interventions: Procedure: different types of ultrasound technique
- Convention ultrasound-guided (Active Comparator): Convention ultrasound-guided biopsy
  Interventions: Procedure: different types of ultrasound technique

INTERVENTIONS:
Procedure: different types of ultrasound technique — Shear-wave elastography-guided or Convention ultrasound-guided

SUMMARY:
To use the shear-wave elastography to assist the transthoracic ultrasound-guided aspiration biopsy of peripheral lung tumor

1. To identify the intra-tumor heterogeneity of elasticity
2. To increase the diagnostic yield in ultrasound-guided transthoracic biopsy of subpleural pulmonary tumor

ELIGIBILITY:
Inclusion criteria:

(1) Patients with radiographic evidence of pulmonary lesions

Exclusion criteria:

1. Age < 20 y/o
2. Patients who cannot hold their breath for 5 seconds
3. Inadequate shear-wave propagation of lung tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield between two groups | 6 months
  sensitivity, specificity, positive predictive value, and negative predictive value

SECONDARY OUTCOMES:
Total times of the biopsy | 1 day
  Total times of the biopsy
Procedure duration | 1 day
  Time duration
Complication rate | 1 day
  Complications like pneumothorax or hemothorax

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) that underlie the results reported in this article, including data dictionaries, will be available upon reasonable request. Additionally, the study protocol, statistical analysis plan, Stata code, and informed consent forms will be shared. Data access will begin three months after publication and remain available for five years. Researchers with methodologically sound proposals may access the data to achieve aims in the approved proposal. Requests for access should be directed to kyw@ntu.edu.tw, and requestors will be required to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data access will begin three months after publication and remain available for five years.
Access Criteria: Researchers with methodologically sound proposals may access the data to achieve aims in the approved proposal.